CLINICAL TRIAL: NCT07031830
Title: APA (Adapted Physical Activity) for Patients With Advanced Melanoma APA (Adapted Physical Activity) for Patients With Advanced Melanoma Undergoing Treatment: Evaluation of a Personalized Program at the Hospital
Brief Title: APA (Adapted Physical Activity) for Patients With Advanced Melanoma
Acronym: APA-M
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0153/OB; N° IDRCB : 2024-A01567-40 (Other: ANSM)
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-12

CONDITIONS: Melanoma of Skin
Keywords: adapted physical activity
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of a personalized program at the hospital through adapted physical activity: Evaluation of a personalized hospital program consisting of 4 months of weekly group sports activity sessions and/or regular in-person and phone motivational interviews for the resumption of physical activity.

SUMMARY:
APA (adapted physical activity) for patients with advanced melanoma APA (adapted physical activity) for patients with advanced melanoma undergoing treatment: evaluation of a personalized program at the hospital Melanoma is a malignant tumor developed from melanocytes. It accounts for approximately 4% of all incident cancers and 1.2% of cancer deaths, regardless of sex.

Since 2011, the advent of new therapies (targeted therapies and immunotherapies) has revolutionized the management of advanced-stage melanoma (unresectable stage III or stage IV).

These treatments have led to a significant improvement in the prognosis of metastatic melanoma, with a 5-year overall survival rate of 34% for targeted therapies, 44% for monotherapy with immunotherapy, and 52% for the combination of nivolumab + ipilimumab.

Due to the improvement in survival rates, advanced melanoma has become a chronic disease affecting all ages. It is therefore essential to maintain the quality of life for these patients.

DETAILED DESCRIPTION:
We know that melanoma and its treatments have an impact on the quality of life of patients: fatigue or impairment of muscular and cardiorespiratory capacities, for example.

Indeed, after a cancer diagnosis, the majority of patients reduce their physical activity. It is estimated that 50 to 75% of these patients do not meet the WHO recommendations (physically inactive). Five years after the cancer diagnosis, nearly half of the patients report limitations in their daily physical activities (walking, carrying, standing for extended periods, etc.).

This physical deconditioning can lead to an exercise intolerance state, resulting in decreased autonomy, quality of life, and self-esteem, along with increased physical and psychological symptoms, and fatigue.

In this context, the High Authority of Health (HAH) has issued several reports integrating physical activity into the care pathway of cancer patients. Indeed, numerous studies have shown the benefits of exercise, particularly in patients with breast or prostate cancer, in order to improve body composition, cardiorespiratory capacity, muscle strength, cancer-related fatigue, pain, anxiety, and quality of life, as well as to prevent treatment-related side effects. Some even mention an impact on survival in prostate cancer.

Currently, despite these reports and various publications illustrating the benefits of physical activity and its feasibility even in metastatic patients, there are many barriers to the prescription of adapted physical activity (APA) by healthcare professionals, who fear, for example, insufficient physical abilities for engaging in sports.

Moreover, to date, few adapted physical activity programs exist in France for patients with advanced melanoma being followed in dermatology. However, this is a population that is sometimes still young and active, requiring the prevention of physical deconditioning and its consequences.

Finally, patients with a history of advanced cancer are sometimes reluctant to resume an activity, Indeed, facing external club partners without health issues, in unfamiliar places, can be a barrier to resuming physical activity. Moreover, patients' motivation wanes over time despite the benefits gained.

Currently, no study has evaluated the interest of a hospital-based adapted physical activity (APA) program consisting of weekly sessions and/or regular in-person and phone motivational interviews for the resumption of physical activity and the maintenance of this activity over time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 or older
* Advanced melanoma treated adjuvantly or curatively with immunotherapy or targeted therapy
* Patient who has read and understood the information letter and does not object to participating in the study
* Member of or beneficiary of a social security scheme
* Patients who have agreed to participate in the adapted sports module

Exclusion Criteria:

* Minor patient
* Melanoma not requiring systemic treatment
* Condition making 6-month follow-up impossible
* Protected incapacitated persons (judicial protection, guardianship, curatorship, deprivation of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced melanoma treated adjuvantly or curatively with immunotherapy or targeted therapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-11-18 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a personalized hospital program | 4 months
  Evaluation of a personalized hospital program consisting of 4 months of weekly collective sports activity sessions for the resumption of physical activity.
Evaluation of a personalized hospital program | 4 months
  Evaluation of a personalized hospital program consisting of 4 months of regular in-person and phone motivational interviews for the resumption of physical activity.

SECONDARY OUTCOMES:
Evaluation of the adherence of patients with advanced melanoma to the physical activity project | 24 months
  Evaluation of the percentage of patients who accepted the sports module (hospital or club) among new patients treated for advanced melanoma during the inclusion period
Evaluation of the maintenance of physical activity over time | 12 months
  Evaluation of - Percentage of patients having maintained physical activity at 12 months according to groups and reason for stopping
Evaluation of the maintenance of physical activity over time | 24 months
  Evaluation of - Percentage of patients having maintained physical activity at 24 months according to groups and reason for stopping
Evaluation of the evolution of physical capacities in the short | At enrollment visit and 6 months
  Assessment of Percentage of improvement in the walking test at enrollment visit
Evaluation of the evolution of physical capacities in the short | "Baseline"
  Assessment of Percentage of improvement in the grip test at enrollment visit
Evaluation of the evolution of physical capacities in the short | "Baseline"
  Assessment of Percentage of improvement in the flexibility test at enrollment visit
Evaluation of the evolution of physical capacities in the short | "Baseline"
  Assessment of Percentage of improvement in the balance test at enrollment visit
Evaluation of the evolution of physical capacities in the long term | 6 months
  Assessment of Percentage of improvement in the walking test between 0 and 6 months
Evaluation of the evolution of physical capacities in the long term | 6 months
  Assessment of Percentage of improvement in the grip test, between 0 and 6 months
Evaluation of the evolution of physical capacities in the long term | 6 months
  Assessment of Percentage of improvement in the flexibility test between 0 and 6 months
Evaluation of the evolution of physical capacities in the long term | 6 months
  Assessment of Percentage of improvement in the balance test between 0 and 6 months
Evaluation of the evolution of quality of life in the short term | "Baseline"
  Evaluation of percentage of improvement in the QLQ C30 score At enrollment visit
Evaluation of the evolution of quality of life in the long term | 6 months, 12 months and 24 months
  Evaluation of percentage of improvement in the QLQ C30 score between 0 and 6 months
Evaluation of the evolution of quality of life in the long term | At enrollment visit, 12 months
  Evaluation of percentage of improvement in the QLQ C30 score 0-12 months
Evaluation of the evolution of quality of life in the long term | At enrollment visit, 24 months
  Evaluation of percentage of improvement in the QLQ C30 score between 0-24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.